CLINICAL TRIAL: NCT03488966
Title: Mindfulness Based Eating Awareness Training (MB-EAT) for Bariatric Surgery Patients: The Effects of Mindfulness on Psychosocial and Physical Functioning
Brief Title: Mindfulness Based Eating Awareness Training for Bariatric Surgery Patients
Acronym: MB-EAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16-5731
Record Dates: First submitted 2017-11-15; First posted 2018-04-05 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Obesity, Morbid; Eating Disorder Symptom
Keywords: Mindfulness; Bariatric Surgery; Obesity; Group psychotherapy
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MB-EAT (Experimental): Behavioral: group psychotherapy. Eight weekly sessions, each session is 2 hours in duration.
  Interventions: Behavioral: Mindfulness Based Eating and Awareness Training
- Waitlist Control (No Intervention): Wait list control.

INTERVENTIONS:
Behavioral: Mindfulness Based Eating and Awareness Training — Eight sessions of Mindfulness Based Eating and Awareness Training (MB-EAT) will be delivered once per week over the course of 8 weeks, following an introductory session. The treatment uses general mindfulness meditation and eating meditation to help participants bring greater awareness and understanding to their relationship with food. Homework consists of weekly mindfulness exercises.
  Arms: MB-EAT

SUMMARY:
The purpose of this study is to evaluate the effects of Mindfulness Based Eating Awareness Training (MB-EAT) for patients who have had bariatric surgery on their weight and mental and physical health compared to patients who do not do this group. All participants will complete questionnaires evaluating eating and mental health before and after the group and 6 and 12 months later. They will have blood pressure readings at these times and complete a questionnaire about their digestive health. Our hypothesis is that participants will maintain their weight loss after bariatric surgery and have improvements in the other outcomes.

DETAILED DESCRIPTION:
MB-EAT may be helpful for reducing emotional eating, overeating and grazing, eating patterns that can lead to weight gain after bariatric surgery. Participants will receive MB-EAT 6 months or more following bariatric surgery. They will be randomly assigned to receive MB-EAT right away or 8 weeks later. Individuals in the group starting in 8 weeks will serve as a waitlist control group.The primary outcome measures will be changes in self-reported eating problems, depression, anxiety, and mindfulness. There will be a follow-up at 6 months and 12 months to establish stability of symptoms post-intervention. Participants will receive one introductory information session about the MB-EAT program, as well as 8 MB-EAT scheduled consecutively over eight weeks. Each session is approximately two hours in length. During MB-EAT, participants will practice mindfulness to help improve their decision making abilities about when and how much to eat. Through MB-EAT, participants will learn to address mindless or out-of-control eating, which can lead to weight gain. Homework will include daily meditations and mindful eating exercises.

ELIGIBILITY:
Inclusion Criteria:

1. Post-bariatric surgery patients recruited from the Toronto Western Hospital-Bariatric Surgery Program (TWH-BSP) who are six months or more post-surgery, are experiencing self-reported difficulties adhering to post-surgery eating guidelines, and can commit to attending the group.
2. Fluent in English.
3. Have the capacity to provide informed consent.

Exclusion Criteria:

1. Active suicidal ideation.
2. Active serious mental illness (i.e., psychotic disorder, bipolar disorder).
3. Active severe depression (i.e., current major depressive disorder diagnosis and PHQ-9 score > 20 [severe depression]).
4. Active severe anxiety (i.e., current anxiety disorder diagnosis and GAD-7 score > 15 [severe anxiety]).
5. Active symptoms of post-traumatic stress disorder (i.e., current diagnosis of post-traumatic stress disorder).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) | Change from baseline to 8 weeks, 6 months, and 12 months
  BMI as calculated by weight (kg) / height (cm)^2
Change in weight | Change from baseline to 8 weeks, 6 months, and 12 months
  Weight in kilograms will be obtained by weighing participants
Height | Baseline
  Height in centimetres will be obtained by measuring participants

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Change from baseline to 8 weeks, 6 months, and 12 months
  A 9-item self-report measure of depression severity that yields a total score. Items are scored from 0-3. Higher values mean more depression. The total score is obtained by summing the items.
Generalized Anxiety Disorder Questionnaire (GAD-7) | Change from baseline to 8 weeks, 6 months, and 12 months
  A 7-item self-report measure of anxiety severity that yields a total score. Items are scored from 0-3. Higher values mean more anxiety. The total score is obtained by summing the items.
The Three Factor Eating Questionnaire -R18 (TFEQ-R18) | Change from baseline to 8 weeks, 6 months, and 12 months
  An 18 item self-report measure of eating behavior that yields a total score. Items are scored from 1-4. Higher values mean more anxiety. The total score is obtained by summing the items.
Five Facets of Mindfulness Questionnaire (FFMQ) | Change from baseline to 8 weeks, 6 months, and 12 months
  A 39-item self-report measuring mindfulness that yields a total score. Items are scored from 1-5. Higher values mean more mindfulness except in the case of the following reverse-scored items: 3, 5, 8, 10, 12, 13, 14, 16, 17, 18, 22, 23, 25, 28, 34, 38, 30, 35, 39. After reverse scoring these items a total score is obtained by summing the items. Average score can be computed by dividing the total score by 39.
Self-Compassion Scale (SCS) | Change from baseline to 8 weeks, 6 months, and 12 months
  A 26-item self-report measure of self-compassion that yields a total score. Items are scored from 1-5. Higher values mean more self-compassion except in the case of the following reverse-scored items: 1, 2, 4, 6, 8, 11, 13, 16, 18, 20, 21, 24, 25. After reverse scoring these items a total score is obtained by summing the items. Average score can be computed by dividing the total score by 26.
Difficulties in Emotion Regulation Scale (DERS) | Change from baseline to 8 weeks, 6 months, and 12 months
  A 36-item self-report questionnaire of emotional difficulties that yields a total score. Items are scored from 1-5. Higher values mean more difficulties in emotion regulation, except in the case of the following reverse-scored items: 1, 2, 6, 7, 8, 10, 17, 20, 22, 24, 34. After reverse scoring these items a total score is obtained by summing the items and an average score is obtained by dividing the sum by 36.
Body Satisfaction Questionnaire (BSQ) | Change from baseline to 8 weeks, 6 months, and 12 months
  A 34-item self-report measure of satisfaction with one's overall body that yields a total score. Items are scored from 0-5. Higher values mean more dissatisfaction with one's body. A total score is obtained by summing the items.
Body Parts Satisfaction Scale (BPSS) | Change from baseline to 8 weeks, 6 months, and 12 months
  An 11-item self-report measure of satisfaction with specific body parts that yields a total score. Items are scored from 0-5. Higher values mean more dissatisfaction. A total score is obtained by summing the items.
The Dichotomous Thinking Scale (DTS) | Change from baseline to 8 weeks, 6 months, and 12 months
  An 11-item self-report scale that measures the cognitive distortions and yields a total score. Items are scored from 1-4 with higher scores indication more cognitive distortions. A total score is obtained by summing the items.
The Obesity Cognitions Scale | Change from baseline to 8 weeks, 6 months, and 12 months
  A 15 item scale that measures cognitive distortions surrounding food, weight, and shape that yields a total score. Items are scored from 0-5 with higher scores indication more cognitive distortions. A total score is obtained by summing the items.
Gastrointestinal Symptom Rating Scale (GSRS) | Change from baseline to 8 weeks, 6 months, and 12 months
  A 15 item self-report scale of gastrointestinal symptoms that yields a total score. Items are scored from 0 to 3 with higher scores indicated more frequent gastrointestinal discomfort. A total score is obtained by summing the items.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Wnuk, Ph.D, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herpertz S, Kielmann R, Wolf AM, Langkafel M, Senf W, Hebebrand J. Does obesity surgery improve psychosocial functioning? A systematic review. Int J Obes Relat Metab Disord. 2003 Nov;27(11):1300-14. doi: 10.1038/sj.ijo.0802410. PMID 14574339
- [Background] Hofmann SG, Sawyer AT, Witt AA, Oh D. The effect of mindfulness-based therapy on anxiety and depression: A meta-analytic review. J Consult Clin Psychol. 2010 Apr;78(2):169-83. doi: 10.1037/a0018555. PMID 20350028
- [Result] Adams CE, Benitez L, Kinsaul J, Apperson McVay M, Barbry A, Thibodeaux A, Copeland AL. Effects of brief mindfulness instructions on reactions to body image stimuli among female smokers: an experimental study. Nicotine Tob Res. 2013 Feb;15(2):376-84. doi: 10.1093/ntr/nts133. Epub 2012 Sep 17. PMID 22987786
- [Result] Alberts HJ, Thewissen R, Raes L. Dealing with problematic eating behaviour. The effects of a mindfulness-based intervention on eating behaviour, food cravings, dichotomous thinking and body image concern. Appetite. 2012 Jun;58(3):847-51. doi: 10.1016/j.appet.2012.01.009. Epub 2012 Jan 10. PMID 22265753
- [Result] Beck NN, Johannsen M, Stoving RK, Mehlsen M, Zachariae R. Do postoperative psychotherapeutic interventions and support groups influence weight loss following bariatric surgery? A systematic review and meta-analysis of randomized and nonrandomized trials. Obes Surg. 2012 Nov;22(11):1790-7. doi: 10.1007/s11695-012-0739-4. PMID 22930073
- [Result] Dalen J, Smith BW, Shelley BM, Sloan AL, Leahigh L, Begay D. Pilot study: Mindful Eating and Living (MEAL): weight, eating behavior, and psychological outcomes associated with a mindfulness-based intervention for people with obesity. Complement Ther Med. 2010 Dec;18(6):260-4. doi: 10.1016/j.ctim.2010.09.008. Epub 2010 Nov 11. PMID 21130363
- [Result] Godsey J. The role of mindfulness based interventions in the treatment of obesity and eating disorders: an integrative review. Complement Ther Med. 2013 Aug;21(4):430-9. doi: 10.1016/j.ctim.2013.06.003. Epub 2013 Jul 9. PMID 23876574
- [Result] Greeson JM. Mindfulness Research Update: 2008. Complement Health Pract Rev. 2009 Jan 1;14(1):10-18. doi: 10.1177/1533210108329862. PMID 20047019
- [Result] Grossman P, Niemann L, Schmidt S, Walach H. Mindfulness-based stress reduction and health benefits. A meta-analysis. J Psychosom Res. 2004 Jul;57(1):35-43. doi: 10.1016/S0022-3999(03)00573-7. PMID 15256293
- [Result] Heatherton TF, Baumeister RF. Binge eating as escape from self-awareness. Psychol Bull. 1991 Jul;110(1):86-108. doi: 10.1037/0033-2909.110.1.86. PMID 1891520
- [Result] Kalarchian MA, Wilson GT, Brolin RE, Bradley L. Binge eating in bariatric surgery patients. Int J Eat Disord. 1998 Jan;23(1):89-92. doi: 10.1002/(sici)1098-108x(199801)23:13.0.co;2-i. PMID 9429923
- [Result] Kristeller JL, Hallett CB. An Exploratory Study of a Meditation-based Intervention for Binge Eating Disorder. J Health Psychol. 1999 May;4(3):357-63. doi: 10.1177/135910539900400305. PMID 22021603
- [Result] Odom J, Zalesin KC, Washington TL, Miller WW, Hakmeh B, Zaremba DL, Altattan M, Balasubramaniam M, Gibbs DS, Krause KR, Chengelis DL, Franklin BA, McCullough PA. Behavioral predictors of weight regain after bariatric surgery. Obes Surg. 2010 Mar;20(3):349-56. doi: 10.1007/s11695-009-9895-6. Epub 2009 Jun 25. PMID 19554382

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT03488966/Prot_SAP_000.pdf